CLINICAL TRIAL: NCT05368844
Title: Harnessing Neurostimulation to Improve Treatment Outcome in Anorexia Nervosa
Brief Title: Transcranial Magnetic Stimulation (TMS) in the Treatment of Anorexia Nervosa
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Guido Frank, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202030
Record Dates: First submitted 2022-04-20; First posted 2022-05-10 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Intervention Model Description: This study aims to test the feasibility, safety and acceptability of a new form of TMS, intermittent theta-burst stimulation (iTBS), in anorexia nervosa and to test whether iTBS can reduce body image distortion and facilitate eating in anorexia nervosa.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active iTBS (Experimental): rTMS treatments will employ the Brainsway stimulator (Brainsway Ltd, Israel). Prior to the first treatment (no more than 5 days prior), each subject's motor threshold (MT) will first be determined according to published methods (Schutter, van Honk, 2006; Julkunen et al, 2009). This location, as well as the stimulation target spot, will be marked at the first session on the scalp and standard methods will be used to target this spot during treatment sessions. The modified BeamF3 scalp heuristic will be used to localize the treatment site over the left DLPFC (Mir-Moghtadaei et al., 2015). Subjects will complete 5 treatments days. A treatment day will consist of 10 treatment sessions with the start of each session timed to be at least 50 minutes from the previous session.
  Interventions: Device: rTMS treatment using BrainsWay Model 104 system with H1-Coil
- Sham iTBS (Sham Comparator): The BrainsWay Model 104 with H4 coil has an integrated sham coil. The sham condition will start with the same clicking noise as the active TMS condition. Every helmet has a corresponding sham H-coil encased in the same helmet. The sham coil induces only a negligible sub-threshold field in the brain while making an identical noise and inducing some scalp sensation. Subjects will complete 5 treatments days. A treatment day will consist of 10 treatment sessions with the start of each session timed to be at least 50 minutes from the previous session. Subjects in this arm will have the option of receiving the Active iTBS protocol after they complete the 5 days of 10 daily treatment sessions.
  Interventions: Device: sham TMS using BrainsWay Model 104 system with H1-Coil

INTERVENTIONS:
Device: rTMS treatment using BrainsWay Model 104 system with H1-Coil — 5 days of 10 daily sessions of rTMS treatment
  Arms: Active iTBS
Device: sham TMS using BrainsWay Model 104 system with H1-Coil — 5 days of 10 daily sessions of sham iTBS treatment
  Arms: Sham iTBS

SUMMARY:
Anorexia nervosa is a severe psychiatric disorder associated with food avoidance and body image distortion, that is feeling fat despite being underweight. It is the third most common chronic illness among adolescent females, and its mortality reaches its peak between the ages 16 and 29 years old. There are very few treatments for anorexia nervosa and especially no biological treatments have been approved. Recent brain imaging research has repeatedly implicated brain circuits that include the insula in the disorder. The insula is a brain region important in taste processing as well as in the integration of body perception and has strong connections to the brain reward system. Transcranial magnetic stimulation (TMS) is a relatively new methodology that has been shown to alter neurocircuitry and alleviate depression. Here, the study goal is to develop TMS as a methodology to change altered neurocircuitry in anorexia nervosa and alleviate disorder specific behaviors.

DETAILED DESCRIPTION:
The goals for this study are 1) to test the feasibility of iTBS in AN and 2) to gather pilot data to as proof of concept of its effectiveness in AN prior to applying for larger funding to the NIH.

Subjects will complete a battery of self-assessments and a diagnostic assessment in order to determine eligibility and for characterization of behavior to be used in later analyses. After eligibility is confirmed, subjects will take part in iTBS treatment over either 1 week (active iTBS groups) or 2 weeks, (1 week sham treatment group, followed by 1 week active iTBS).

The design will be a randomized control design that also includes a cross over design. Subjects will be randomized to either Group 1, Active iTBS, or Group 2, Sham/Active iTBS.

Group 1 will receive active iTBS over 5 days, with 10 brief sessions per day (5 study days/50 session total). Group 2 will receive Sham over 5 days, with 10 brief sessions per day, and this will be followed by active iTBS over 5 days, with 10 brief sessions per day (20 study days/100 session total).

ELIGIBILITY:
Inclusion Criteria:

* Females ages 18 to 45 years
* Diagnostic criteria. Current diagnosis of AN according to the DSM V, including having a severe fear of weight gain and body image distortion
* Restricting or binge/purge subtype
* English is primary language spoken

Exclusion Criteria:

* Subjects who are pregnant or think they may be pregnant will be excluded from the study.
* Subjects will not have electrolyte, blood count or kidney or liver function abnormalities. Prior to starting the TMS treatment (Visit 2), all subjects will complete a basic metabolic panel (must be completed within no more than one week prior to the start of the TMS treatment) to rule out electrolyte or metabolic abnormalities.
* Subjects may not have a lifetime history of a condition likely to be associated with increased intracranial pressure, space occupying brain lesion, any history of seizure except those therapeutically induced by ECT or a febrile seizure of infancy or single seizure related to a known drug related event.
* Subjects may not have a history of significant head trauma with loss of consciousness for greater than 5 minutes.
* Subjects may not have an intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed.
* Subjects may not currently take more than lorazepam 2 mg daily (or equivalent) or any dose of an anticonvulsant due to the potential to limit TMS efficacy or have a history of lack of response to accelerated course of iTBS or rTMS in the past.
* Subjects may not have a concomitant major unstable medical illness, cardiac pacemaker or implanted medication pump.
* Subjects may not have symptoms of alcohol or substance abuse or dependence in the past month, may not have previous or current organic brain syndromes, psychotic disorders, bipolar type disorders, somatization disorders, or conversion disorder.
* Antidepressant bupropion or other seizure threshold lowering medication or are currently taking tricyclic antidepressants or neuroleptics.
* Permanent eye makeup (such as eyeliner or eyebrows) or other face tattoos due to potential ferrous materials used in the tattoo ink
* Subjects may not have a history of neurocardiogenic syncope as there is an increased risk of TMS-induced neurocardiogenic syncope in adolescent populations.
* Subjects may not have implanted neurostimulators, intracardiac lines, or heart disease that causes moderate to severe symptoms and/or is characterized by moderate to severe pathology (including a recent history of myocardial infarction and heart failure with an ejection fraction of less than 30% or with a New York Heart Association Functional Classification of Class III or IV).
* Subjects may not have a history of stroke or other brain lesions.
* Subjects may not have a history of suicide attempt(s).
* Subject may not have a family history of epilepsy.
* Cannot refrain from drinking alcohol for the duration of the study. Subjects will be asked to refrain from consuming alcohol for the duration of the study. At the beginning of each treatment day subjects will be asked about alcohol consumption in the last 48 hours and will not complete the treatment sessions that day if they have had alcohol in the last 48 hours.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-06-16 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of TMS sessions | at study completion, up to 2 weeks
  To establish feasibility of iTBS in anorexia nervosa the investigator will assess the following: total percent of sessions completed by the subject.
Acceptability of TMS procedures | at study completion, up to 2 weeks
  To establish acceptability of iTBS in anorexia nervosa the investigator will assess the following: subjects will be asked open-ended questions about the subject's experience of the study.

SECONDARY OUTCOMES:
Eating Disorders Inventory 3 Drive for Thinness Subscale | Change from baseline to study completion, up to 2 weeks
  The Eating Disorders Inventory 3 is a self report assessment that measures core eating disorder symptoms. Subjects will complete this measure at the beginning and end of the study and the investigator will measure the change in scores. The Drive for Thinness Subscale has a range of 0 to 28 where higher scores mean worse outcome.
Eating Disorders Inventory 3 (EDI-3) Body Dissatisfaction Subscale | Change from baseline to study completion, up to 2 weeks
  The Eating Disorders Inventory 3 is a self report assessment that measures core eating disorder symptoms. Subjects will complete this measure at the beginning and end of the study and the investigator will measure the change in scores. The Drive for Thinness Subscale has a range of 0 to 40 where higher scores mean worse outcome.
Weight gain | Change in body mass index from baseline to study completion, up to 2 weeks
  Body Mass Index over time as a measure of food intake from the start to end of the study.
Spielberger State-Trait Anxiety Scale-Version Y (STAI-Y) State Anxiety Subscale | Change from baseline to study completion, up to 2 weeks
  The Spielberger State-Trait Anxiety Scale-Version Y is a self report assessment that measure state and trait anxiety. Subjects will complete this measure at the beginning and end of the study and the investigator will measure the change in scores of State Anxiety. State anxiety has a range of 0 to 80 with higher scores indicating worse outcome.
Spielberger State-Trait Anxiety Scale-Version Y (STAI-Y) Trait Anxiety Subscale | Change from baseline to study completion, up to 2 weeks
  The Spielberger State-Trait Anxiety Scale-Version Y is a self report assessment that measure state and trait anxiety. Subjects will complete this measure at the beginning and end of the study and the investigator will measure the change in scores of Trait Anxiety. Trait anxiety has a range of 0 to 80 with higher scores indicating worse outcome.
Beck Depression Inventory | Change from baseline to study completion, up to 2 weeks
  The Beck Depression Inventory is a self report assessment that measures depression. Subjects will complete this measure at the beginning and end of the study and the investigator will measure the change in scores. The score range is from 0 to 63 with higher scores indicating worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Guido Frank, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cole EJ, Stimpson KH, Bentzley BS, Gulser M, Cherian K, Tischler C, Nejad R, Pankow H, Choi E, Aaron H, Espil FM, Pannu J, Xiao X, Duvio D, Solvason HB, Hawkins J, Guerra A, Jo B, Raj KS, Phillips AL, Barmak F, Bishop JH, Coetzee JP, DeBattista C, Keller J, Schatzberg AF, Sudheimer KD, Williams NR. Stanford Accelerated Intelligent Neuromodulation Therapy for Treatment-Resistant Depression. Am J Psychiatry. 2020 Aug 1;177(8):716-726. doi: 10.1176/appi.ajp.2019.19070720. Epub 2020 Apr 7. PMID 32252538
- [Background] Schutter DJ, van Honk J. A standardized motor threshold estimation procedure for transcranial magnetic stimulation research. J ECT. 2006 Sep;22(3):176-8. doi: 10.1097/01.yct.0000235924.60364.27. PMID 16957532
- [Background] Mir-Moghtadaei A, Caballero R, Fried P, Fox MD, Lee K, Giacobbe P, Daskalakis ZJ, Blumberger DM, Downar J. Concordance Between BeamF3 and MRI-neuronavigated Target Sites for Repetitive Transcranial Magnetic Stimulation of the Left Dorsolateral Prefrontal Cortex. Brain Stimul. 2015 Sep-Oct;8(5):965-73. doi: 10.1016/j.brs.2015.05.008. Epub 2015 May 29. PMID 26115776
- [Background] Frank GKW, DeGuzman MC, Shott ME. Motivation to eat and not to eat - The psycho-biological conflict in anorexia nervosa. Physiol Behav. 2019 Jul 1;206:185-190. doi: 10.1016/j.physbeh.2019.04.007. Epub 2019 Apr 10. PMID 30980856